CLINICAL TRIAL: NCT00467038
Title: Treatment of Aggression, Anger and Emotional Dysregulation in Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDA-2-038-06F
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2015-08-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Borderline Personality Disorder
Keywords: affect; aggression; anger; behavior therapy; borderline personality disorder; MRI, functional
MeSH Terms: conditions — Borderline Personality Disorder; Aggression | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dialectical Behavior Therapy (Other): Dialectical Behavior Therapy
  Interventions: Behavioral: Dialectical Behavior
- Healthy Controls (No Intervention): Healthy controls

INTERVENTIONS:
Behavioral: Dialectical Behavior — Dialectical Behavior Therapy is an empirically validated treatment approach emphasizing the role of emotion regulation in the treatment of suicidal and self-destructive behaviors in BPD
  Arms: Dialectical Behavior Therapy

SUMMARY:
This study examines the effects of 12 months of dialectical behavior therapy (DBT) for subjects with borderline personality disorder on aggression, anger and emotional dysregulation. Treatment effects will be measured by changes in interview, self-report, psychophysiology testing and fMRI neuroimaging.

DETAILED DESCRIPTION:
Borderline Personality Disorder (BPD) is a disabling disorder characterized by poor affect regulation and poor impulse control. This often results in impaired interpersonal relationships and maladaptive behavioral patterns, including anger dyscontrol, aggression towards others and self-destructive behaviors. Evidence suggests that is a relatively common disorder, affecting 2% of the population 1. In addition, BPD patients have more frequent psychiatric hospitalizations, greater use of outpatient psychotherapy and more visits to the emergency room than individuals with any other psychiatric disorder 3, 4. Due to the heterogeneity of symptoms that fall under the DSM-IV definition of BPD, the most productive efforts to understand the underlying neurobiology of this disorder have employed a dimensional approach. This application focuses on the domain of affective instability and altered emotion regulation, believed by many to be at the core of the disorder 5.

The emotional dysregulation of BPD appears to be a biological vulnerability. This vulnerability includes both increased emotional reactivity, as well as an impaired capacity to employ effortful control in the modulation of emotional reactions. The emotional reactivity is manifested by high sensitivity to emotional stimuli and heightened emotional intensity5 and may reflect limbic system over activity. The impairment in emotional modulation results in a slow return to the baseline emotional state and may reflect deficits in prefrontal regulatory regions. While data supporting this formulation are limited, self-report measures of responses to various emotional stimuli and more recently, objective, non-verbal physiological measures including startle eye blink modulation (SEM), have been used to test this theory.

SEM is a well-established technique used to study the psychophysiology of emotion and has been shown to reflect amygdala activation6. Our research group has demonstrated exaggerated affective startle in BPD patients compared to healthy control subjects at later probe positions in response to words with emotionally negative valence, selected specifically to target emotions commonly unpleasant for BPD patients. Emerging neurobiological theories based on preliminary functional neuroimaging studies posit that BPD is a hyperarousal-dyscontrol syndrome 4, implicating dysfunction in amygdala activity coupled with weakening of prefrontal inhibitory control. Several neuroimaging studies from our research group have helped advance this idea7. Building on these exciting findings and the expertise available, this project uses a translational approach to study treatment effects on emotional regulation in BPD with SEM and prediction of treatment response with functional magnetic resonance imaging (fMRI).

Dialectical Behavior Therapy is an empirically validated treatment approach emphasizing the role of emotion regulation in the treatment of suicidal and self-destructive behaviors in BPD8, 9. It has gained considerable popularity and is included as a component of the APA guidelines for treatment of BPD10. While this approach stresses skills and techniques for emotional regulation, and encourages cognitive control over maladaptive behavioral patterns, there have been neither neuroimaging nor psychophysiological studies of the effect of DBT on emotional processing in BPD, despite its proven efficacy. While neuroimaging and psychophysiological studies of a psychotherapeutic treatment have been done in major depression 11, 12 13, no such studies have been done in BPD. By examining changes in affective startle and baseline predictors of response with fMRI blood oxygenation level dependent (BOLD) activation patterns associated with DBT treatment, this project aims to better characterize the nature of emotional dysregulation in BPD, and identify features that predict a good response to DBT treatment. In addition, the project will explore the relationship between clinical improvement of BPD symptomatology with DBT treatment and changes in neurobiological measures by performing follow-up SEM after six and twelve months of DBT treatment. This approach will help elucidate the neuroanatomy of abnormal emotional processing in BPD and may help identify potential strategies for correcting these deficits.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* In good physical health as confirmed by a complete physical exam, electrocardiogram, neurological exam, and routine laboratory tests of blood and urine
* A negative urine toxicology screen
* Completion of psychiatric evaluations, medical evaluations, and self-report questionnaires through separate protocol- Biological Correlates of Personality Disorders (GCO #88-244)

  1. meet DSM-IV criteria for borderline personality disorder and have an overt aggression scale- modified aggression subscale score of six or above on one of two OASM pre-treatment screens.
  2. not currently be taking any psychiatric medications. If they have taken psychiatric medications in the past, they must be at least 2 weeks (6 half-lives) medication-free prior to participating in the study. These medications include mood stabilizers, antidepressants, antipsychotics, and benzodiazepines.

Exclusion Criteria:

* meet criteria for schizophrenia, bipolar I disorder, schizoaffective disorder or any other psychotic disorder.
* have met criteria for substance abuse or dependence during the 6 months prior to entry into the study
* have a past history of intravenous drug use, cocaine abuse or dependence, or any substance dependence that resulted in serious medical sequelae
* meet criteria for current MDE, as they may require antidepressant treatment
* have made a suicide attempt or had a psychiatric hospitalization during the 6 months prior to entry into the study
* be on any psychotropic medication(s) upon entry into the study
* be in concurrent psychotherapy (case management services and work therapy programs are not considered individual psychotherapy)
* be pregnant or lactating

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2006-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Goodman, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States

REFERENCES:
- [Result] Goodman M, Carpenter D, Tang CY, Goldstein KE, Avedon J, Fernandez N, Mascitelli KA, Blair NJ, New AS, Triebwasser J, Siever LJ, Hazlett EA. Dialectical behavior therapy alters emotion regulation and amygdala activity in patients with borderline personality disorder. J Psychiatr Res. 2014 Oct;57:108-16. doi: 10.1016/j.jpsychires.2014.06.020. Epub 2014 Jul 2. PMID 25038629

RESULTS

PARTICIPANT FLOW:
Groups:
- Dialectical Behavior Therapy: Participants receiving Dialectical Behavior Therapy
- Healthy Controls: Healthy controls- no intervention
Period: Overall Study
Arm/Group | Dialectical Behavior Therapy | Healthy Controls
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dialectical Behavior Therapy: Dialectical Behavior Therapy
  Dialectical Behavior: Dialectical Behavior Therapy is an empirically validated treatment approach emphasizing the role of emotion regulation in the treatment of suicidal and self-destructive behaviors in BPD
  Event-related fMRI was obtained pre- and post-12-months of standard-DBT in unmedicatedBPD patients.
- Healthy Controls: Healthy controls
  Age and gender matched healthy volunteers
- Total: Total of all reporting groups
Arm/Group | Dialectical Behavior Therapy | Healthy Controls | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (11.5) | 30.4 (10.4) | 31.6 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Self-Report of Difficulties in Emotion Regulation (DERS)
Description: The present study examines DBT treatment effect on emotion regulation in unmedicated outpatients with BPD as measured by changes in the Difficulties in Emotion Regulation Scale. The DERS is a brief, 36-item, self-report questionnaire.
  DERS total score ranges from 36- 180. Higher scores reflect higher difficulties in emotion regulation.
  The measure yields a total score as well as scores on six scales derived through factor analysis:
  1. Nonacceptance of emotional responses, 2. Difficulties engaging in goal directed behavior, 3. Impulse control difficulties, 4. Lack of emotional awareness, 5. Limited access to emotion regulation strategies, 6. Lack of emotional clarity Responses are on a 5-point scale: 1=almost never, 2=sometimes, 3=about half the time, 4=most of the time, 5=almost always
Time Frame: 12 months
Population: 22 age- and gender-matched unmedicated BPD and HC participants (11 in each group).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Healthy Controls: Healthy controls age- and gender-matched to other group of participants
Arm/Group | Dialectical Behavior Therapy | Healthy Controls
Number analyzed (Participants) | 11 | 11
units on a scale
  12 month | 101.5 (25.7) | 54.8 (14.4)
  Baseline | 120.5 (24.2) | 56.6 (14.9)
Statistical Analysis 1: Comparison: Dialectical Behavior Therapy vs Healthy Controls; Test type: Superiority or Other; p < 0.004, t-test, 1 sided; <0.004 p value was common for all time points

2. Secondary Outcome: Group x Time Interaction Amygdala Activity
Description: 0 to 12 month difference scores in group x time interaction amygdala activity
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: bold signal units
Groups:
- Dialectical Behavior Therapy: Dialectical Behavior Therapy is an empirically validated treatment approach emphasizing the role of emotion regulation in the treatment of suicidal and self-destructive behaviors in BPD
Arm/Group | Dialectical Behavior Therapy | Healthy Controls
Number analyzed (Participants) | 11 | 11
bold signal units | -11.54 (11.73) | 16.67 (1.99)
Statistical Analysis 1: Comparison: Dialectical Behavior Therapy vs Healthy Controls; Test type: Superiority or Other; p = 0.08, Fisher's LSD post-hoc, trend level

ADVERSE EVENTS:
Time Frame: 4 years, between 2007 and 2010
Groups:
- Arm 1: Dialectical Behavior Therapy
  Dialectical Behavior: Dialectical Behavior Therapy is an empirically validated treatment approach emphasizing the role of emotion regulation in the treatment of suicidal and self-destructive behaviors in BPD
- Arm 2: Healthy controls- no intervention
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/11
Other Adverse Events (participants affected / at risk) | 7/11 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=11) | Arm 2 (N=11)
Psychiatric hospitalization after suicidal ideation and unsafe behavior (Psychiatric disorders) | 1 | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=11) | Arm 2 (N=11)
Vertebrae fracture due to fall (General disorders) | 1 | 0
Arrest due to armed robbery (Social circumstances) | 1 | 0
Excessive drinking and unsafe sex (General disorders) | 1 | 0
Superficial cut as deliberate self-harm (Psychiatric disorders) | 1 | 0
Superficial scratching as deliberate self-harm (Psychiatric disorders) | 1 | 0
Treatment for eating disorder (Psychiatric disorders) | 1 | 0
Anxiety and dizziness during fMRI scan (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Small community sample. Additionally, our emotional task was a "passive viewing task" which means that we did not examine "active" emotion regulation, per se which might be considered a study limitation by some. No comparison treatment group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes